CLINICAL TRIAL: NCT03918031
Title: Personalized Feedback for Distress Intolerant Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brooke Kauffman, Principal Investigator, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000686; 1F31DA046127-01 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-04-17 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Anxiety Disorders; Depression; Psychological Distress; Tobacco Dependence; Smoking, Tobacco; Smoking, Cigarette
Keywords: Psychological Distress; Tobacco; Smoking; Feedback; Stress; Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression; Tobacco Use Disorder; Tobacco Smoking; Cigarette Smoking; Smoking | interventions — Smoking Devices

STUDY DESIGN:
Intervention Model Description: If participant meets eligibility criteria, the participant will be randomly assigned to complete a one-session computer-delivered intervention: either (1) personalized feedback intervention on ability to handle discomfort and smoking or (2) personalized feedback intervention on smoking only.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFI for Smoking & Distress Tolerance (Active Comparator): A brief, one-session computer-delivered personalized feedback intervention (PFI) that addresses smoking and distress tolerance.
  Interventions: Behavioral: PFI for Smoking & Distress Tolerance
- PFI for Smoking Only (Active Comparator): A brief, one-session computer-delivered personalized feedback intervention (PFI) that addresses smoking only (no distress tolerance component).
  Interventions: Behavioral: PFI for Smoking Only

INTERVENTIONS:
Behavioral: PFI for Smoking & Distress Tolerance — Personalized Feedback Intervention for smoking and distress tolerance.
  Arms: PFI for Smoking & Distress Tolerance
Behavioral: PFI for Smoking Only — Personalized Feedback Intervention for smoking only (no distress tolerance component)
  Arms: PFI for Smoking Only

SUMMARY:
This project will develop and refine a computer-delivered integrated Personalized Feedback Intervention (PFI) that directly addresses smoking and distress tolerance. The PFI will focus on feedback about smoking behavior, distress tolerance, and adaptive coping strategies.

DETAILED DESCRIPTION:
The primary goal of the research study is to investigate the efficacy of a brief, personalized computer-delivered transdiagnostic intervention (PFI) that addresses smoking and distress tolerance to reduce smoking, increase quit attempts, reduce perceived barriers to cessation, increase distress tolerance, reduce anxiety/depressive symptoms, and increase adaptive coping skills compared to a personalized feedback on smoking only control. To address this aim, the investigators will implement a randomized controlled trial that will employ a longitudinal experimental design and involve four stages: (a) phone-screener (pre-screener); (b) baseline appointment consisting of a pre-intervention assessment (eligibility), random assignment to a one-session computer-delivered intervention (Active PFI versus Control PFI with no personalized feedback on distress tolerance), and a post-intervention assessment; (c) 2-week follow-up; (d) 1-month follow-up. Assessments will include a multi-method approach, including biological, behavioral, and self-report methods.

ELIGIBILITY:
Inclusion Criteria:

* Low distress tolerance defined as a DTS mean score of 2.56 or lower
* Daily smoking for at least one year (minimum 5 cigarettes per day and biochemically confirmed via Carbon Monoxide [CO] analysis at least 5 ppm)

Exclusion Criteria:

* Currently engaging in treatment for an alcohol/drug problem including smoking cessation
* Legal status that will interfere with participating
* Not being fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Kauffman, M.A., Principal Investigator — University of Houston; Michael Zvolensky, Ph.D., Principal Investigator — University of Houston
Locations (1):
- Anxiety and Health Research Laboratory and Substance Use Treatment Clinic, University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project Website — https://www.uh.edu/class/psychology/clinical-psych/research/restore/projects/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
Started | 57 | 64
Post-Intervention | 57 | 64
2-Week Follow-up | 57 | 60
1-Month Follow-up | 56 | 62
Completed | 57 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only | Total
Number analyzed (Participants) | 57 | 64 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.60 (5.35) | 29.98 (9.01) | 29.33 (7.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 39 | 47 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 17 | 23 | 40
  White | 39 | 32 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 64 | 121
Timeline Follow-Back [Mean (Standard Deviation); unit: cigarettes/day] | 8.26 (2.98) | 8.64 (2.53) | 8.46 (2.75)

OUTCOME MEASURES:

1. Primary Outcome: Rulers for Smoking Cessation
Description: The Rulers for Smoking Cessation asks participants to rate three rulers associated with motivation, confidence, and intention to quit smoking. Motivation is indexed by, "How important is stopping smoking to you (0 = Not important at all; 10 = Most important goal of my life)?" with a higher score indicating a better outcome. Confidence is indexed by, "How confident are you that you will quit smoking within the next month (0 = Not at all; 10 = 100% confident)?" with a higher score indicating a better outcome. Intention is indexed by, "How ready are you to quit smoking within the next month (0 = Not at all; 10 = 100% ready)?" with a higher score indicating a better outcome.
Time Frame: Baseline, 2-week, and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
Number analyzed (Participants) | 57 | 64
units on a scale
  Motivation to Quit: Baseline | 7.37 (2.57) | 7.89 (2.05)
  Motivation to Quit: 2-Week Follow-up: number analyzed (Participants) | 57 | 60
  Motivation to Quit: 2-Week Follow-up | 8.58 (1.46) | 8.40 (1.71)
  Motivation to Quit: 1-Month Follow-up: number analyzed (Participants) | 56 | 62
  Motivation to Quit: 1-Month Follow-up | 8.39 (1.46) | 7.98 (2.32)
  Confidence to Quit: Baseline | 6.09 (2.81) | 6.48 (2.39)
  Confidence to Quit: 2-Week Follow-up: number analyzed (Participants) | 57 | 60
  Confidence to Quit: 2-Week Follow-up | 8.09 (2.26) | 7.78 (2.18)
  Confidence to Quit: 1-Month Follow-up: number analyzed (Participants) | 56 | 62
  Confidence to Quit: 1-Month Follow-up | 8.02 (1.81) | 7.73 (2.34)
  Intention to Quit: Baseline | 6.53 (2.87) | 7.20 (2.61)
  Intention to Quit: 2-Week Follow-up: number analyzed (Participants) | 57 | 60
  Intention to Quit: 2-Week Follow-up | 7.98 (2.44) | 7.95 (2.22)
  Intention to Quit: 1-Month Follow-up: number analyzed (Participants) | 56 | 62
  Intention to Quit: 1-Month Follow-up | 8.34 (1.54) | 7.66 (2.52)

2. Primary Outcome: Barriers to Cessation Scale
Description: The Barriers to Cessation Scale assesses 19-barriers, or specific stressors, associated with smoking cessation. Participants indicate, according to a 4-point Likert-style scale (0 = Not a barrier to 3 = Large barrier), the extent to which they identify with each of the barriers to cessation. Lower scores indicate a better outcome (range = 0 - 57).
Time Frame: Baseline, 2-week, and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
Number analyzed (Participants) | 57 | 64
score on a scale
  Baseline | 38.46 (8.20) | 38.61 (9.01)
  2-Week Follow-up: number analyzed (Participants) | 57 | 60
  2-Week Follow-up | 32.67 (9.95) | 33.08 (11.09)
  1-Month Follow-up: number analyzed (Participants) | 56 | 62
  1-Month Follow-up | 31.23 (9.90) | 31.18 (12.13)

3. Primary Outcome: Timeline Follow-Back
Description: The Timeline Follow-Back (TLFB) is a self-report measure to assess retrospective estimates of daily smoking. The TLFB was used to assess smoking rate computed as a mean score of past 7-day cigarettes smoked per day.
Time Frame: Baseline, 2-week, and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
Number analyzed (Participants) | 57 | 64
cigarettes/day
  Baseline | 8.26 (2.98) | 8.64 (2.53)
  2-Week Follow-up: number analyzed (Participants) | 57 | 60
  2-Week Follow-up | 4.19 (3.21) | 4.26 (3.05)
  1-Month Follow-up: number analyzed (Participants) | 56 | 62
  1-Month Follow-up | 3.12 (3.10) | 3.06 (3.19)

4. Primary Outcome: Distress Tolerance Scale
Description: The Distress Tolerance Scale is a self-report measure in which respondents indicate, on a 5-point Likert-type scale (1 = 'strongly agree' to 5 = 'strongly disagree'), the extent to which they believe they can experience and withstand distressing emotional states. All items are averaged to create a total mean score ranging from 1 to 5 with higher total scores indicating a better outcome (i.e., greater tolerance for distress).
Time Frame: Baseline, 2-week, and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
Number analyzed (Participants) | 57 | 64
score on a scale
  Baseline | 1.69 (0.38) | 1.75 (0.44)
  2-Week Follow-up: number analyzed (Participants) | 57 | 60
  2-Week Follow-up | 2.51 (0.75) | 2.57 (0.73)
  1-Month Follow-up: number analyzed (Participants) | 56 | 62
  1-Month Follow-up | 2.76 (0.82) | 2.72 (0.89)

5. Primary Outcome: Mood and Anxiety Symptom Questionnaire-Short Form
Description: The Mood and Anxiety Symptom Questionnaire-Short Form will be used to assess anxiety/depressive symptoms. Participants indicate how much they have experienced each symptom on a 5-point Likert-type scale (1 = Not at all to 5 = Extremely). Specifically, the Anxious Arousal subscale will be used to measure anxiety and the Anhedonic Depression subscale will be used to measure depression. The Anxious Arousal subscale consists of 17-items with lower scores indicating better outcomes (range = 17 - 85). The Anhedonic Depression subscale consists of 22-items with lower scores indicating better outcomes (range = 22 - 110).
Time Frame: Baseline, 2-week, and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
Number analyzed (Participants) | 57 | 64
score on a scale
  Anxiety: Baseline | 54.14 (18.73) | 51.40 (19.51)
  Anxiety: 2-Week Follow-up: number analyzed (Participants) | 57 | 60
  Anxiety: 2-Week Follow-up | 44.12 (17.80) | 43.07 (19.18)
  Anxiety: 4-Week Follow-up: number analyzed (Participants) | 56 | 62
  Anxiety: 4-Week Follow-up | 41.75 (18.78) | 42.55 (20.35)
  Depression: Baseline | 71.26 (14.67) | 70.05 (12.29)
  Depression: 2-Week Follow-up: number analyzed (Participants) | 57 | 60
  Depression: 2-Week Follow-up | 62.30 (9.89) | 60.97 (14.50)
  Depression: 4-Week Follow-up: number analyzed (Participants) | 56 | 62
  Depression: 4-Week Follow-up | 58.18 (12.33) | 59.74 (15.33)

6. Primary Outcome: Self-Help Scale
Description: The Self-Help Scale asks participants to indicate whether they would be willing to try each of 10 strategies to help deal with depression and anxiety on a 5-point Likert-type scale from 0 (definitely not) to 4 (extremely willing). Higher scores indicate a better outcome (range = 0 - 4).
Time Frame: Baseline, 2-week, and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
Number analyzed (Participants) | 57 | 64
score on a scale
  Baseline | 3.00 (0.76) | 3.00 (0.72)
  2-Week Follow-up: number analyzed (Participants) | 57 | 60
  2-Week Follow-up | 3.09 (0.76) | 2.96 (0.77)
  1-Month Follow-up: number analyzed (Participants) | 56 | 62
  1-Month Follow-up | 3.23 (0.66) | 3.01 (0.72)

ADVERSE EVENTS:
Time Frame: 1-month
Arm/Group | PFI for Smoking & Distress Tolerance | PFI for Smoking Only
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/64
Other Adverse Events (participants affected / at risk) | 0/57 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03918031/Prot_SAP_001.pdf